CLINICAL TRIAL: NCT06454734
Title: Lower Limb Lymphedema Treatment by Extracorporeal Shock Wave Therapy: Clinical Trial
Brief Title: Shock Wave Therapy for Lower Limb Lymphedema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Roser Belmonte, Rehabilitation specialist, MD, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023/11201/I
Record Dates: First submitted 2024-05-28; First posted 2024-06-12 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Lymphedema, Lower Limb
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Intervention Model Description: Double blind randomized clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients, outcome assessors and investigators will not know if received treatment was placebo or therapeutic. The physiotherapist will apply the treatment according to a list of random numbers generated to make 2 treatment groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DLT + ESWT (Experimental): To DLT + ESWT group, decongestive lymphatic therapy (DLT) plus radial extracorporeal wave treatment (ESWT) will be applied, at a dose and intensity probed to be useful to diminish volume in upper limb lymphedema.
  Interventions: Device: Extracorporeal shock wave therapy by radial device; Other: DLT
- DLT + Sham ESWT (Sham Comparator): To DLT + Sham ESWT group, decongestive lymphatic therapy plus sham radial extracorporeal wave treatment will be applied, at a placebo dose and intensity.
  Interventions: Device: Placebo extracorporeal shock wave therapy by radial device; Other: DLT

INTERVENTIONS:
Device: Extracorporeal shock wave therapy by radial device — Patients will receive treatment by extracorporeal shock waves therapy (ESWT).
  Other Names: Radial ESWT; rESWT
  Arms: DLT + ESWT
Device: Placebo extracorporeal shock wave therapy by radial device — Patients will receive treatment sham extracorporeal shock waves.
  Other Names: Radial ESWT; rESWT
  Arms: DLT + Sham ESWT
Other: DLT — Patients will receive treatment with decongestive lymphatic therapy (DLT: manual lymphatic drainage, compression)
  Other Names: Decongestive Lymphatic Therapy

SUMMARY:
This is a double-blind randomized clinical trial to compare the effect of shock wave therapy on lower limb lymphedema. There are two arms: A) complex decongestive therapy + extracorporeal shock waves therapy; B) complex decongestive therapy plus placebo extracorporeal shock waves.

DETAILED DESCRIPTION:
This is a double blind, randomized, clinical trial. 30 patients with lower limb lymphedema will be randomized in 2 groups. One group will receive the habitual complex decongestive therapy (lymphatic manual drainage and compression) plus extracorporeal shock waves therapy. The other group will receive complex decongestive therapy (lymphatic manual drainage and compression) plus placebo extracorporeal shock waves.

Patients in the 2 groups will be instructed on skin care measures and kinesitherapy. The usual manual lymphatic drainage and compression will be applied to the 2 groups. The 2 groups will receive 10 treatment sessions, 2 weekly for 5 weeks.

Group complex decongestive therapy + shock waves. Patients will receive treatment with manual lymphatic drainage, compression, and shock waves.

Group complex decongestant therapy + placebo. Patients will receive treatment with manual lymphatic drainage, compression, and placebo shock waves.

Tolerance and possible adverse effects will be recorded by physiotherapist. Any adverse effect detected will be evaluated by the rehabilitation medical doctor.

ELIGIBILITY:
Inclusion criteria

* Patients with lower limb lymphedema
* Lymphedema of at least 6 months of evolution
* The lymphedema must affect at least the knee to the foot
* Moderate or severe lymphedema (grades 2 or 3)
* Sign the informed consent

Exclusion criteria

* Under 18 years of age
* Coagulation disorders (hemophilia, treatment with acenocoumarol, etc.)
* Current or previous deep vein thrombosis of the lower extremity
* Pregnancy
* Electronic implantable medical devices as pacemaker implants, medication pumps, etc
* Having received treatment with complex decongestive therapy or shock waves during the last 6 months
* Treatment with corticosteroids or radiotherapy in the area to be treated in the last 6 weeks
* Active oncological disease in the area to be treated
* Active infectious-inflammatory process in the area to be treated
* Cognitive or sensory deficits that prevent collaboration
* Inability to walk independently or inability to attend therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Limb volume change 1 | 5 weeks
  The difference between limb volume previous of treatment and at the end of treatment

SECONDARY OUTCOMES:
Limb volume change 2 | 9 weeks
  The difference between limb volume from previous of treatment to 1 month after
VAS Pain | 9 weeks
  Changes in pain at previous treatment, at the end of treatment and to 1 month after. Measured by a visual analogue scale (VAS) (from 0 not pain to 10 maximum imaginable)
VAS Heaviness | 9 weeks
  Changes in heaviness from previous treatment, to the end of treatment and to 1 month after. Measured by a visual analogue scale (VAS) (from 0 not heaviness to 10 maximum imaginable)
VAS Hardness | 9 weeks
  Changes in hardness from previous treatment, to the end of treatment and to 1 month after. Measured by a visual analogue scale (VAS) (from 0 not hardness to 10 maximum imaginable)

OTHER OUTCOMES:
Water composition | 9 weeks
  Changes in water lower limb composition at previous treatment, to the end of treatment anto 1 month after.

CONTACTS AND LOCATIONS:
Overall Officials: Roser Belmonte, MD, PhD, Principal Investigator — Hospital del Mar
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rankin J, Morris K, Reilly A. The All-Ireland Guidelines for the diagnosis, assessment and management of lymphoedema. Br J Community Nurs. 2022 Oct 1;27(Sup10):S22-S26. doi: 10.12968/bjcn.2022.27.Sup10.S22. PMID 36205409
- [Background] Bae H, Kim HJ. Clinical outcomes of extracorporeal shock wave therapy in patients with secondary lymphedema: a pilot study. Ann Rehabil Med. 2013 Apr;37(2):229-34. doi: 10.5535/arm.2013.37.2.229. Epub 2013 Apr 30. PMID 23705118
- [Background] Tsai YL, I TJ, Chuang YC, Cheng YY, Lee YC. Extracorporeal Shock Wave Therapy Combined with Complex Decongestive Therapy in Patients with Breast Cancer-Related Lymphedema: A Systemic Review and Meta-Analysis. J Clin Med. 2021 Dec 19;10(24):5970. doi: 10.3390/jcm10245970. PMID 34945266
- [Background] Lee KW, Kim SB, Lee JH, Kim YS. Effects of Extracorporeal Shockwave Therapy on Improvements in Lymphedema, Quality of Life, and Fibrous Tissue in Breast Cancer-Related Lymphedema. Ann Rehabil Med. 2020 Oct;44(5):386-392. doi: 10.5535/arm.19213. Epub 2020 Sep 28. PMID 32986941